CLINICAL TRIAL: NCT02166905
Title: A Phase I/IIb Study of DEC205mAb-NY-ESO-1 Fusion Protein (CDX-1401) Given With Adjuvant Poly-ICLC in Combination With INCB024360 for Patients in Remission With Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma Whose Tumors Express NY-ESO-1 or LAGE-1 Antigen
Brief Title: DEC-205/NY-ESO-1 Fusion Protein CDX-1401, Poly ICLC, and IDO1 Inhibitor INCB024360 in Treating Patients With Ovarian, Fallopian Tube, or Primary Peritoneal Cancer in Remission
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Celldex Therapeutics (Industry); Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 248613; NCI-2014-00771 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 248613 (Other: Roswell Park Cancer Institute); P30CA016056 (NIH)
Record Dates: First submitted 2014-04-21; First posted 2014-06-18 (Estimated); Results first posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-01

CONDITIONS: Fallopian Tube Carcinoma; Ovarian Carcinoma; Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — epacadostat; poly ICLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (CDX-1401, poly ICLC) (Experimental): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 and poly ICLC as in Phase I.
  Interventions: Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Poly ICLC
- Arm II (CDX-1401, poly ICLC, IDO1 inhibitor INCB024360) (Experimental): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401, poly ICLC, and IDO1 inhibitor INCB024360 as in Phase I.
  Interventions: Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401; Drug: Epacadostat; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Poly ICLC

INTERVENTIONS:
Biological: DEC-205/NY-ESO-1 Fusion Protein CDX-1401 — Given via intracutaneous injection
  Other Names: CDX-1401
Drug: Epacadostat — Given PO
  Other Names: INCB 024360; INCB024360
  Arms: Arm II (CDX-1401, poly ICLC, IDO1 inhibitor INCB024360)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Poly ICLC — Given SC
  Other Names: Hiltonol; Poly I:Poly C with Poly-L-Lysine Stabilizer; poly-ICLC; PolyI:PolyC with Poly-L-Lysine Stabilizer; Polyinosinic-Polycytidylic Acid Stabilized with Polylysine and Carboxymethylcellulose; Polyriboinosinic-Polyribocytidylic Acid-Polylysine Carboxymethylcellulose; Stabilized Polyriboinosinic/Polyribocytidylic Acid

SUMMARY:
This partially randomized phase I/IIb trial studies the side effects and best dose of IDO1 inhibitor INCB024360 in combination with DEC-205/NY-ESO-1 fusion protein CDX-1401 and poly ICLC and to see how well they work in treating patients with ovarian, fallopian tube, or primary peritoneal cancer who no longer have evidence of disease. Antigens (such as cancer/testis antigen [NY-ESO-1] protein) are found on many cancer cells. Vaccines made from NY-ESO-1 protein may cause the immune system to produce immune cells and antibodies that may help locate the NY-ESO-1 and/or cancer/testis antigen 2 (LAGE-1) antigens on cancer cells. By finding them, the immune system may then work to control or eliminate the remaining cancer cells. INCB024360 is an inhibitor of an enzyme called indoleamine 2,3 dioxygenase (IDO). This enzyme is produced by tumor cells to disable immune cells, and limit the efficacy of immune attack. Giving DEC-205/NY-ESO-1 fusion protein CDX-1401 with poly ICLC and IDO1 inhibitor INCB024360 may generate stronger and more long lasting anti-cancer immune responses in patients with ovarian, fallopian tube, and primary peritoneal cancer in remission.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of fixed doses of DEC205mAb-NY-ESO-1 fusion protein (DEC-205/NY-ESO-1 fusion protein CDX-1401) with adjuvant poly-ICLC given as a vaccine in combination with INCB024360 (IDO1 inhibitor INCB024360). (Phase I) II. To evaluate toxicity as defined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0. (Phase I) III. To determine the progression free survival (PFS) (primary endpoint) using standard immune-related response criteria (irRC) criteria. (Phase IIb)

SECONDARY OBJECTIVES:

I. To determine the effectiveness of INCB024360 on enhancing vaccine efficacy by assessing cancer-testis antigen (NY-ESO-1) specific cellular and humoral immunity.

II. To determine the effectiveness of Sirolimus on enhancing vaccine efficacy by assessing NY-ESO-1 specific cellular and humoral immunity (Exploratory Cohort ONLY) III. Peripheral blood NY-ESO-1 specific cluster of differentiation (CD)8+ and CD4+ T cells. (Exploratory Cohort ONLY) IV. Peripheral blood NY-ESO-1 specific antibodies.(Exploratory Cohort ONLY) V. Peripheral blood frequency of CD4+CD25+forkhead box P3 (FOXP3)+ regulatory T cells. (Exploratory Cohort ONLY) VI. Pharmacokinetics of INCB02360 in relation to T cell frequency and function in correlation with PFS. (Exploratory Cohort ONLY)

OUTLINE:

PHASE I:

Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 via intracutaneous injection on day 1, poly ICLC subcutaneously (SC) on days 1 and 2, and IDO1 inhibitor INCB024360 orally (PO) twice daily (BID) on days 1-28. Treatment repeats every 28 days for up to 5 courses in the absence of disease progression or unacceptable toxicity. Patients receive IDO1 inhibitor INCB024360 for up to 7 courses.

PHASE IIb: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401 and poly ICLC as in Phase I.

ARM II: Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401, poly ICLC, and IDO1 inhibitor INCB024360 as in Phase I.

After completion of study treatment, patients are followed up for 30 days and then at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients will be women with epithelial ovarian, fallopian tube, or primary peritoneal carcinoma after chemotherapy with no evidence of disease or minimal residual disease for primary or recurrent disease; this may or may not be measurable; these patients would normally enter a period of observation after standard management
* Any human leukocyte antigen (HLA) type; (historic HLA typing is permitted)
* Tumor expression of NY-ESO-1 or LAGE-1 by immunohistochemistry (IHC) and/or reverse transcriptase polymerase chain reaction (RTPCR)
* Life expectancy > 6 months
* Absolute neutrophil count (ANC) >= 1,000/uL
* Platelets (PLT) >= 100,000/uL
* Hemoglobin (Hgb) >= 8 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Serum aspartate aminotransferase (serum glutamic oxaloacetic transaminase [SGOT]/AST) or serum alanine aminotransferase (serum glutamate pyruvate transaminase [SGPT]/ALT) =< 3 x ULN
* Serum creatinine =< 2 x ULN
* Have been informed of other treatment options
* Patient or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* The ability to swallow and retain oral medication
* Patients of child-bearing potential must agree to use acceptable contraceptive methods (e.g., double barrier) during treatment
* Patients may have received previous NY-ESO-1 vaccine therapy; patients who received maintenance paclitaxel or bevacizumab are eligible for enrollment provided they have discontinued therapy (at least 4 weeks for prior taxane or prior bevacizumab) prior to randomization and recovered from toxicities to less than grade 2

Exclusion Criteria:

* Metastatic disease to the central nervous system for which other therapeutic options, including radiotherapy, may be available
* Other serious illnesses (e.g., serious infections requiring antibiotics, bleeding disorders)
* History of severe autoimmune disorders requiring use of steroids or other immunosuppressives
* Concomitant systemic treatment with chronic use (based on the investigator's judgment) of corticosteroids, anti-histamine or non-steroidal anti-inflammatory drugs, and other platelet inhibitory agents
* Chemotherapy, radiation therapy, or immunotherapy within 4 weeks prior to first dosing of study drug (6 weeks for nitrosoureas); concomitant hormonal therapies for breast cancers are allowed
* Subjects being treated with a monoamine oxidase inhibitor (MAOI), or drug which has significant MAOI activity (e.g., Meperidine, linezolid, methylene blue) within 3 weeks prior to screening
* Subjects who are currently receiving therapy with a potent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inducer or inhibitor (e.g. clarithromycin, telithromycin, nefazodone, itraconazole, ketoconazole, atazanavir)
* Use of UDP glucuronosyltransferase 1 family, polypeptide A9 (UGT1A9) inhibitor including: diclofenac, imipramine, and ketoconazole
* Participation in any other clinical trial involving another investigational agent within 4 weeks prior to first dosing of study drug
* Known hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* Mental impairment that may compromise the ability to give informed consent and comply with the requirements of the study
* Lack of availability of a patient for immunological and clinical follow-up assessment
* Evidence of current drug or alcohol abuse or psychiatric impairment, which in the Investigator's opinion will prevent completion of the protocol therapy or follow-up
* Pregnant or nursing female patients
* Unwilling or unable to follow protocol requirements
* Any condition which in the Investigator's opinion deems the patient an unsuitable candidate to receive study drug (i.e., any significant medical illness or abnormal laboratory finding that would, in the investigator's judgment, increase the patient's risk by participating in this study)
* Known hypersensitivity to any of the study drugs that will be given to the participant
* Additional exclusion criteria for exploratory cohort ONLY: Known pulmonary hypertension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-10-10 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emese Zsiros, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I (CDX-1401, Poly ICLC); Phase IIb arm2 (CDX-1401, Poly ICLC, With IDO1 Inhibitor INCB024360): DEC205mAb-NY-ESO-1 fusion protein (1 mg,intracutaneous injection) on Day 1 of each 28 day cycle for a total of 5 cycles.
  Adjuvant poly-ICLC (1 ml, subcutaneous) on Day 1 and Day 2 of each 28 day cycle for a total of 5 cycles
  + INCB024360 (Oral) : 300 mg BID for a total of 7 cycles
- Phase IIb arm1 (CDX-1401, Poly ICLC, IDO1 Without Inhibitor INCB024360): DEC205mAb-NY-ESO-1 fusion protein (1 mg,intracutaneous injection) on Day 1 of each 28 day cycle for a total of 5 cycles.
  Adjuvant poly-ICLC (1 ml, subcutaneous) on Day 1 and Day 2 of each 28 day cycle for a total of 5 cycles
- Phase IIb Arm 3 (Exploratory Cohort. Enrollment at Roswell Park Site ONLY. ): DEC205mAb-NY-ESO-1 fusion protein (1 mg,intracutaneous injection) on Day 1 of each 28 day cycle for a total of 5 cycles.
  Adjuvant poly-ICLC (1 ml, subcutaneous) on Day 1 and Day 2 of each 28 day cycle for a total of 5 cycles
  + Sirolimus: 4 cycles of 4 mg/day for 2 weeks followed by 2 weeks off
Period: Overall Study
Arm/Group | Phase I (CDX-1401, Poly ICLC) | Phase IIb arm1 (CDX-1401, Poly ICLC, IDO1 Without Inhibitor INCB024360) | Phase IIb arm2 (CDX-1401, Poly ICLC, With IDO1 Inhibitor INCB024360) | Phase IIb Arm 3 (Exploratory Cohort. Enrollment at Roswell Park Site ONLY. )
Started | 7 | 16 | 15 | 2
Completed | 6 | 16 | 15 | 2
Not Completed | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Eligible patients will be women ≥ 18 years, with epithelial ovarian, fallopian tube, or primary peritoneal carcinoma after chemotherapy with no evidence of disease or minimal residual disease for primary or recurrent disease.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I (CDX-1401, Poly ICLC) | Phase IIb arm1 (CDX-1401, Poly ICLC, IDO1 Without Inhibitor INCB024360) | Phase IIb arm2 (CDX-1401, Poly ICLC, With IDO1 Inhibitor INCB024360) | Phase IIb Arm 3 (Exploratory Cohort. Enrollment at Roswell Park Site ONLY. ) | Total
Number analyzed (Participants) | 6 | 16 | 15 | 2 | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 10 | 11 | 1 | 26
  >=65 years | 2 | 6 | 4 | 1 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (12) | 65 (10) | 63 (10) | 63 (8) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 16 | 15 | 2 | 39
  Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 16 | 14 | 2 | 38
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Safety and Evaluate Toxicity of Fixed Doses for Phase I Patients
Description: To determine the safety of fixed doses of DEC205mAb-NY-ESO-1 fusion protein with adjuvant poly-ICLC given as a vaccine in combination with INCB024360 300mg, number of Participants with Dose Limiting Toxicities is reported
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Phase I (CDX-1401, Poly ICLC, and a Fixed Daily Dose of INCB024360 ): Patients will receive a fixed intracutaneous dose of DEC205mAb-NY-ESO-1 fusion protein (CDX-1401) (Day 1) given with subcutaneous adjuvant poly-ICLC (Day 1 and Day 2) for each 28 day cycle for a total of 5 cycles; and Cohort 1 patient enrollment will begin INCB024360 at a fixed daily dose (300mg ) of BID orally
Arm/Group | Phase I (CDX-1401, Poly ICLC, and a Fixed Daily Dose of INCB024360 )
Number analyzed (Participants) | 6
Participants | 1

2. Primary Outcome: Progression Free Survival (PFS) Based on Immune Related Response Criteria (irRC) for Phase II Patients
Description: Percentage of Participants with Progression Free Survival Using irRC Criteria for Phase II Patients are reported. irRC criteria disease progression is defined as at least 25% increase in tumor burden compared with nadir (at any single time point) in two consecutive observations at least 4 weeks apart.
Time Frame: Up to 6 months
Population: Progression free survival rates (proportion) at 6 months are reported.
Measure: Number (90% Confidence Interval); unit: Proportion of participants w/o Progress
Arm/Group | Phase IIb arm1 (CDX-1401, Poly ICLC, IDO1 Without Inhibitor INCB024360) | Phase IIb arm2 (CDX-1401, Poly ICLC, With IDO1 Inhibitor INCB024360) | Phase IIb Arm 3 (Exploratory Cohort. Enrollment at Roswell Park Site ONLY. )
Number analyzed (Participants) | 16 | 15 | 2
Proportion of participants w/o Progress | 0.78 [0.52 to 0.91] | 0.54 [0.29 to 0.73] | 0.50 [0.02 to 0.88]
Statistical Analysis 1: Comparison: Phase IIb arm1 (CDX-1401, Poly ICLC, IDO1 Without Inhibitor INCB024360); Test type: Other; p = 0.177, Log Rank; Hazard Ratio (HR) = 0.4, 90% CI 2-sided [0.1 to 1.2] — Reference=arm 1

3. Primary Outcome: To Evaluate Toxicity as Defined by NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Description: All patients enrolled in this study will be eligible for the analysis of toxicity. The toxicity rate will be estimated using a one-sided, 95%, exact binomial confidence interval (Clopper-Pearson).
Time Frame: Up to 12 months
Measure: Number; unit: participants
Groups:
- Phase I (CDX-1401, Poly ICLC, and a Fixed Daily Dose of INCB024360 ): Patients will receive a fixed intracutaneous dose of DEC205mAb-NY-ESO-1 fusion protein (CDX-1401) (Day 1) given with subcutaneous adjuvant poly-ICLC (Day 1 and Day 2) for each 28 day cycle for a total of 5 cycles; and Cohort 1 patient enrollment will begin INCB024360 at a fixed daily dose of BID orally
- Arm II 2a (CDX-1401, Poly ICLC, Without IDO1 Inhibitor INCB024360): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401, poly ICLC, without IDO1 inhibitor INCB024360 in phase IIb.
  DEC-205/NY-ESO-1 Fusion Protein CDX-1401: Given via intracutaneous injection
  Epacadostat: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Poly ICLC: Given SC
- Arm II 2b (CDX-1401, Poly ICLC, With IDO1 Inhibitor INCB024360): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401, poly ICLC, with IDO1 inhibitor INCB024360 in phase IIb.
  DEC-205/NY-ESO-1 Fusion Protein CDX-1401: Given via intracutaneous injection
  Epacadostat: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Poly ICLC: Given SC
- Phase IIb Arm 3 (Exploratory Cohort ): 4 cycles of sirolimus in combination with DEC205mAb-NY-ESO-01 fusion protein (CDX-1401) with adjuvant poly-ICLC
Arm/Group | Phase I (CDX-1401, Poly ICLC, and a Fixed Daily Dose of INCB024360 ) | Arm II 2a (CDX-1401, Poly ICLC, Without IDO1 Inhibitor INCB024360) | Arm II 2b (CDX-1401, Poly ICLC, With IDO1 Inhibitor INCB024360) | Phase IIb Arm 3 (Exploratory Cohort )
Number analyzed (Participants) | 6 | 16 | 15 | 2
participants
  Serious Adverse Events | 2 | 1 | 2 | 0
  Other Adverse Events | 6 | 14 | 15 | 2

4. Secondary Outcome: Antibody Titers
Description: Due to the PI leaving the institute, these biomarker data were not generated and are therefore not available to be analyzed.
Time Frame: Up to 12 months
Population: There were 0 patients with this information analyzed. All efforts were made to retrieve data.
Arm/Group | Phase I (CDX-1401, Poly ICLC, and a Fixed Daily Dose of INCB024360 ) | Arm II 2a (CDX-1401, Poly ICLC, Without IDO1 Inhibitor INCB024360) | Arm II 2b (CDX-1401, Poly ICLC, With IDO1 Inhibitor INCB024360) | Phase IIb Arm 3 (Exploratory Cohort )
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Frequency of Memory T Cell Populations
Description: as for outcome 4
Time Frame: Up to 12 months
Population: There were 0 patients with this information analyzed. All efforts were made to retrieve data.
Arm/Group | Phase I (CDX-1401, Poly ICLC, and a Fixed Daily Dose of INCB024360 ) | Arm II 2a (CDX-1401, Poly ICLC, Without IDO1 Inhibitor INCB024360) | Arm II 2b (CDX-1401, Poly ICLC, With IDO1 Inhibitor INCB024360) | Phase IIb Arm 3 (Exploratory Cohort )
Number analyzed (Participants) | 0 | 0 | 0 | 0

6. Secondary Outcome: NY-ESO-1 Specific CD8+ and CD4+ Frequency and Function
Description: as for outcome 4
Time Frame: Up to 12 months
Population: There were 0 patients with this information analyzed. All efforts were made to retrieve data.
Arm/Group | Phase I (CDX-1401, Poly ICLC, and a Fixed Daily Dose of INCB024360 ) | Arm II 2a (CDX-1401, Poly ICLC, Without IDO1 Inhibitor INCB024360) | Arm II 2b (CDX-1401, Poly ICLC, With IDO1 Inhibitor INCB024360) | Phase IIb Arm 3 (Exploratory Cohort )
Number analyzed (Participants) | 0 | 0 | 0 | 0

7. Secondary Outcome: T Cell Receptor (TCR) Avidity
Description: as for outcome 4
Time Frame: Up to 12 months
Population: There were 0 patients with this information analyzed. All efforts were made to retrieve data.
Arm/Group | Phase I (CDX-1401, Poly ICLC, and a Fixed Daily Dose of INCB024360 ) | Arm II 2a (CDX-1401, Poly ICLC, Without IDO1 Inhibitor INCB024360) | Arm II 2b (CDX-1401, Poly ICLC, With IDO1 Inhibitor INCB024360) | Phase IIb Arm 3 (Exploratory Cohort )
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Between the start date of intervention until 30 days after the last intervention or until the study participant is lost to follow up, the start of new treatment, or until the study investigator assesses the event(s) as stable or irreversible, up to 1 year.
Groups:
- Phase II 2a (CDX-1401, Poly ICLC): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401, poly ICLC, without IDO1 inhibitor INCB024360 in phase IIb.
  DEC-205/NY-ESO-1 Fusion Protein CDX-1401: Given via intracutaneous injection
  Epacadostat: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Poly ICLC: Given SC
- Phase II 2b (CDX-1401, Poly ICLC With INCB024360): Patients receive DEC-205/NY-ESO-1 fusion protein CDX-1401, poly ICLC, with IDO1 inhibitor INCB024360 in phase IIb.
  DEC-205/NY-ESO-1 Fusion Protein CDX-1401: Given via intracutaneous injection
  Epacadostat: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Pharmacological Study: Correlative studies
  Poly ICLC: Given SC
- Phase II 3 (Exploratory Cohort): 4 cycles of sirolimus in combination with DEC205mAb-NY-ESO-01 fusion protein (CDX-1401) with adjuvant poly-ICLC
Arm/Group | Phase I (CDX-1401, Poly ICLC, and a Fixed Daily Dose of INCB024360 ) | Phase II 2a (CDX-1401, Poly ICLC) | Phase II 2b (CDX-1401, Poly ICLC With INCB024360) | Phase II 3 (Exploratory Cohort)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/16 | 3/15 | 0/2
Serious Adverse Events (participants affected / at risk) | 2/6 | 1/16 | 2/15 | 0/2
Other Adverse Events (participants affected / at risk) | 6/6 | 14/16 | 15/15 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (CDX-1401, Poly ICLC, and a Fixed Daily Dose of INCB024360 ) (N=6) | Phase II 2a (CDX-1401, Poly ICLC) (N=16) | Phase II 2b (CDX-1401, Poly ICLC With INCB024360) (N=15) | Phase II 3 (Exploratory Cohort) (N=2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (CDX-1401, Poly ICLC, and a Fixed Daily Dose of INCB024360 ) (N=6) | Phase II 2a (CDX-1401, Poly ICLC) (N=16) | Phase II 2b (CDX-1401, Poly ICLC With INCB024360) (N=15) | Phase II 3 (Exploratory Cohort) (N=2)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 3 (3) | 3 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (4) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 3 (5) | 1 (1) | 2 (2) | 0 (0)
Early satiety (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (4) | 3 (3) | 6 (8) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 4 (5) | 6 (7) | 2 (2)
Injection site discolouration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 6 (11) | 6 (6) | 7 (7) | 0 (0)
Injection site nodule (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 4 (11) | 4 (5) | 4 (4) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 2 (7) | 4 (6) | 1 (1)
Injection site swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splinter (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carbon dioxide increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombosis in device (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 4 (5) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/05/NCT02166905/Prot_SAP_000.pdf